CLINICAL TRIAL: NCT05032937
Title: Clinical Study of Domestic Polysaccharide Superparamagnetic Iron Oxide Nanoparticle Injection for Coronary Artery Contrast-enhanced Magnetic Resonance Contrast-enhanced Angiography
Brief Title: the Accuracy and Safety of Coronary Artery Contrast-enhanced Magnetic Resonance Imaging With Polysaccharide Superparamagnetic Iron Oxide Nanoparticle
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Chunjian Li, Dr., MD, Ph.D, Director of CCU Ward, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 012
Record Dates: First submitted 2021-08-21; First posted 2021-09-02 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Coronary Heart Disease
Keywords: Ultrasmall Superparamagnetic Particles of Iron Oxide; Contrast-Enhanced Magnetic Resonance; Plaque Stability
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ECMR (Experimental): Patients will receive contrast-enhanced cardiac magnetic resonance with polysaccharide superparamagnetic iron oxide nanoparticle before percutaneous coronary angiography.
  Interventions: Drug: domestic polysaccharide superparamagnetic iron oxide nanoparticle

INTERVENTIONS:
Drug: domestic polysaccharide superparamagnetic iron oxide nanoparticle — Patients will receive contrast-enhanced cardiac magnetic resonance with polysaccharide superparamagnetic iron oxide nanoparticle before percutaneous coronary angiography.Patients received intravenous polysaccharide superparamagnetic iron oxide nanoparticle before magnetic resonance imaging.

SUMMARY:
This is a single-center, prospective, controlled and diagnostic clinical trial which will enroll 30 patients scheduled for coronary angiography in China.Patients will receive contrast-enhanced cardiac magnetic resonance with polysaccharide superparamagnetic iron oxide nanoparticle before percutaneous coronary angiography.In order to evaluate the safety of polysaccharide superparamagnetic iron oxide nanoparticle, patients will detect iron levels in peripheral and tissue before and after the examination.The main indicators of the study are the degree of coronary artery stenosis and the stability of coronary atherosclerotic plaque assessed by contrast-enhanced cardiac magnetic resonance with polysaccharide superparamagnetic iron oxide nanoparticle.

ELIGIBILITY:
Inclusion Criteria:

* Age ≧ 18 years, < 75 years;
* Patients who planned coronary angiography ;
* Patients with normal renal function or CKD stage 1-3;
* Patients themselves or authorized families to sign informed consent voluntarily.

Exclusion Criteria:

* Patients who were allergic to iodine contrast agent or had allergic history or allergic constitution to iron and dextran;
* Patients who can ' t accept magnetic resonance examination because of psychological ( such as autism syndrome ) or physical reasons ( such as metal retention in the body );
* Malignancies or other comorbid conditions with life expectancy less than 1 year;
* Pregnant or lactating woman;
* Hearing impaired persons;
* Cardiac function grade III-IV;
* History of coronary stenting or coronary artery bypass grafting;
* Patients who were taking other iron agents orally or intravenously;
* Patients with hemosiderin deposition or hemochromatosis;
* Patients with acute coronary syndromes;
* Any other patients that researcher deems it's unsuitable to be admitted.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
The degree of coronary artery stenosis | baseline
  Degree of coronary artery stenosis assessed by contrast-enhanced cardiac magnetic resonance with polysaccharide superparamagnetic iron oxide nanoparticle.
The degree of coronary artery stenosis | 72 hours
  Degree of coronary artery stenosis assessed by quantitative coronary angiography.
Plaque stability of coronary atherosclerotic plaques | baseline
  Plaque stability of coronary atherosclerotic plaques assessed by contrast-enhanced cardiac magnetic resonance with polysaccharide superparamagnetic iron oxide nanoparticle.
Plaque stability of coronary atherosclerotic plaques | 72 hours
  Plaque stability of coronary atherosclerotic plaques assessed by Optical coherence tomography.
Blood routine | baseline,72 hours,30 Days,3 months
  Blood routine examination of patients before and after examination to evaluate general condition of patients.
Blood biochemistry | baseline,72 hours,30 Days,3 months
  Blood biochemistry examination of patients before and after examination to evaluate liver function.
Urine routine | baseline,72 hours,30 Days,3 months
  Urine routine examination of patients before and after examination to evaluate kidney function.
24-hour urine biochemistry | baseline,72 hours,30 Days,3 months
  24-hour urine biochemistry examination of patients before and after examination to evaluate kidney function.
Retinol binding protein | baseline,72 hours,30 Days,3 months
  Retinol binding protein examination of patients before and after examination to evaluate kidney function.
Neutrophil gelatinase-associated lipocalin | baseline,72 hours,30 Days,3 months
  Neutrophil gelatinase-associated lipocalin examination of patients before and after examination to evaluate kidney function.
Serum iron | baseline,72 hours,30 Days,3 months
  Determination of serum iron before and after ECMR to evaluate the changes of iron content in peripheral blood.
Ferritin | baseline,72 hours,30 Days,3 months
  Determination of serum ferritin before and after ECMR to evaluate the changes of iron content in peripheral blood.
Transferrin | baseline,72 hours,30 Days,3 months
  Determination of serum transferrin before and after ECMR to evaluate the changes of iron content in peripheral blood.
Change of iron content in tissues between different time points | baseline,6 months
  Evaluation of tissue iron content by T1W MRI before and after ECMR.

CONTACTS AND LOCATIONS:
Overall Officials: Chunjian Li, Dr, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dong Z, Si G, Zhu X, Li C, Hua R, Teng J, Zhang W, Xu L, Qian W, Liu B, Wang J, Wang T, Tang Y, Zhao Y, Gong X, Tao Z, Xu Z, Li Y, Chen B, Kong X, Xu Y, Gu N, Li C. Diagnostic Performance and Safety of a Novel Ferumoxytol-Enhanced Coronary Magnetic Resonance Angiography. Circ Cardiovasc Imaging. 2023 Jul;16(7):580-590. doi: 10.1161/CIRCIMAGING.123.015404. Epub 2023 Jul 18. PMID 37463240
- [Derived] Kar A, Gupta S, Matilal A, Kumar D, Sarkar S. Nanotherapeutics for the Myocardium: A Potential Alternative for Treating Cardiac Diseases. J Cardiovasc Pharmacol. 2023 Sep 1;82(3):180-188. doi: 10.1097/FJC.0000000000001444. PMID 37341530